CLINICAL TRIAL: NCT04467671
Title: Prospective, Open-labeled, Single-arm Clinical Trial to Evaluate the Safety and Efficacy of the Second-generation Tissue Engineered Vascular Graft as Vascular Conduits for Extracardiac Total Cavopulmonary Connection.
Brief Title: Two-Year Study of the Safety and Efficacy of the Second-Generation Tissue Engineered Vascular Grafts
Acronym: TEVG-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Gunze Limited (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE18703; 5UH3HL148693 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: HLH - Hypoplastic Left Heart Syndrome; DORV; DILV - Double Inlet Left Ventricle; Mitral Atresia; Tricuspid Atresia; Unbalanced AV Canal; Single-ventricle; Heart Defects, Congenital; Cardiovascular Abnormalities; Cardiovascular Diseases; Heart Diseases
Keywords: Fontan; TEVG; Tissue Engineered Vascular Graft
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tricuspid Atresia; Univentricular Heart; Heart Defects, Congenital; Cardiovascular Abnormalities; Cardiovascular Diseases; Heart Diseases | interventions — Blood Vessel Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Tissue Engineered Vascular Grafts (Experimental)
  Interventions: Combination Product: Tissue Engineered Vascular Grafts

INTERVENTIONS:
Combination Product: Tissue Engineered Vascular Grafts — Patients will undergo EC TCPC interposition grafting with a tissue engineered vascular graft and serial magnetic resonance imaging (MRI)

SUMMARY:
A single arm clinical trial evaluating the safety and efficacy of the second generation TEVG as vascular conduits for extracardiac total cavopulmonary connection.

DETAILED DESCRIPTION:
This investigation is a prospective, open-labeled clinical trial determining the safety of the use of tissue engineered vascular grafts as conduits for EC TCPC. Patients will be monitored for adverse events (AE) and serious adverse events (SAE). Special attention will be paid to the incidence of stenosis. We will determine graft-related morbidity and mortality for the second generation TEVGs which will include any post-operative complication such as any aneurismal dilation, stenosis, thromboembolic or infectious event that requires treatment and is thought to be caused by the graft as determined by the investigators and confirmed by the data safety monitoring board. The graft related complication rates will be compared between the first and second generation TEVGs. An interim analysis will be performed to assess the incidence of early (<6 month) graft-related complications in the first 6 enrolled patients. Safety and tolerability will be assessed through serial imaging, to determine the effect of growth and remodeling on graft performance through echocardiography and 4-dimensional MRI. All appropriate patients requiring EC TCPC who meet study inclusion/exclusion criteria will be evaluated for enrollment in the clinical trial. All enrolled subjects will be required to have follow-up visits at Nationwide Children's Hospital for a minimum of 2 years following implant. After obtaining informed consent for the patient's parents, patients with single ventricle cardiac anomalies will undergo EC TCPC using a tissue engineered conduit. Post-operative care and monitoring will follow an established, standardized, clinical algorithm in which the patient's clinical status including complications and measurements of graft function will be serially evaluated and recorded over a two year period using physical examination, echocardiography, and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in the study if they meet all of the following criteria.

  1. Patient must be a candidate to undergo an extracardiac total cavopulmonary connection.
  2. Patient and/or legal guardian must voluntarily provide informed consent/assent for participation in the study.

Exclusion Criteria:

* Patients will be excluded from participation in the study if they meet any of the following criteria.

  1. Patient has an urgent/emergent operative status.
  2. Patient has acute renal failure or renal insufficiency in the opinion of the investigator
  3. Patient requires a graft less than 12 mm or greater than 24 mm in diameter.
  4. Patient has a pacemaker.
  5. Patient has pulmonary vascular resistance greater than 4 um2 (u=Wood's units)
  6. Patient has abnormal venous drainage (interrupted inferior vena cava [IVC]).
  7. Patient presents with significant atrio-ventricular valve regurgitation that in the opinion of the investigator, makes them ineligible.
  8. Patient has a history of another condition or significant medical problem that, in the opinion of the investigator, precludes compliance with protocol-specified procedures.
  9. Patients taking any medications that in the opinion of the Investigator could interfere with the TEVG, including bisphosphonates (i.e. Clodronate or Zoledronate).
  10. Patient or parent/legal guardian is, in the opinion of the investigator, unable to comply with protocol evaluations.
  11. Preoperative hemoglobin <11.0 mg/dL at time of patient's pre-admission testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of TEVG | 2 years
  Assessed through graft related complications as determined by serial echocardiogram
Safety and Tolerability of TEVG | 2 years
  Assessed through graft related complications as determined by serial MRI
Safety and Tolerability of TEVG | 2 years
  Assessed through adverse events

SECONDARY OUTCOMES:
Efficacy of TEVG | 2 years
  Evaluate graft performance based on MRI
Efficacy of TEVG | 2 years
  Measured graft volume(mL) as determined by MRI
Efficacy of TEVG | 2 years
  Measured graft length (mm) as determined by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Breuer, MD, Study Chair — Nationwide Children's Hospital; Toshiharu Shinoka, MD/PhD, Study Chair — Nationwide Children's Hospital; Mark Galantowicz, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Biological Samples: We plan to make available representative samples of the bone marrow-derived mononuclear cells and seeded scaffold to a NIH-designated entity (RM Innovation Catalyst) for in depth and independent characterization. Specifically, for each TEVG manufactured, 1 ml of bone marrow-derived mononuclear cells and a 5mm x 5mm section of the seeded scaffold will be sampled, packed, and transported to the RM Innovation Catalyst per their instructions. In addition, copies of the batch record and completed certificate of analysis will be forwarded to the NIH-designated laboratory.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Prior to study initiation, the US FDA will have a comprehensive description of the processes followed to assure the accuracy, reliability, integrity, availability, and authenticity of required records and signatures supporting the data reported in the CSR will be provided to the Agency for confirmation that it will support a regulatory filing for TEVG. Every 6 months throughout the study, data will be shared with RM Innovation Catalyst, with a final locked data set no later than six months prior to the end of the award. Data from our long-term follow up policy will be made available on an annual basis if requested by the RM Innovation Catalyst or the NIH.
Access Criteria: De-identified data will be provided to RM Innovation Catalyst. A Clinical Study Report will be submitted to the US FDA following the International Conference on Harmonization E3 Guideline for Industry: Structure and Content of Clinical Study Reports. Summary results of the trial will be submitted to ClinicalTrial.gov within one year of the primary completion date (per regulation and NIH policy). Results of screening tests and subjects participation in the study and ongoing test results will be shared with their primary care physician and/or primary cardiologist if cardiac care is being provided outside of Nationwide Children's Hospital.

REFERENCES:
- [Background] Drews JD, Pepper VK, Best CA, Szafron JM, Cheatham JP, Yates AR, Hor KN, Zbinden JC, Chang YC, Mirhaidari GJM, Ramachandra AB, Miyamoto S, Blum KM, Onwuka EA, Zakko J, Kelly J, Cheatham SL, King N, Reinhardt JW, Sugiura T, Miyachi H, Matsuzaki Y, Breuer J, Heuer ED, West TA, Shoji T, Berman D, Boe BA, Asnes J, Galantowicz M, Matsumura G, Hibino N, Marsden AL, Pober JS, Humphrey JD, Shinoka T, Breuer CK. Spontaneous reversal of stenosis in tissue-engineered vascular grafts. Sci Transl Med. 2020 Apr 1;12(537):eaax6919. doi: 10.1126/scitranslmed.aax6919. PMID 32238576
- [Background] Ruiz-Rosado JD, Lee YU, Mahler N, Yi T, Robledo-Avila F, Martinez-Saucedo D, Lee AY, Shoji T, Heuer E, Yates AR, Pober JS, Shinoka T, Partida-Sanchez S, Breuer CK. Angiotensin II receptor I blockade prevents stenosis of tissue engineered vascular grafts. FASEB J. 2018 Jun 15;32(12):fj201800458. doi: 10.1096/fj.201800458. Online ahead of print. PMID 29906242
- [Background] Lee YU, Mahler N, Best CA, Tara S, Sugiura T, Lee AY, Yi T, Hibino N, Shinoka T, Breuer C. Rational design of an improved tissue-engineered vascular graft: determining the optimal cell dose and incubation time. Regen Med. 2016 Mar;11(2):159-67. doi: 10.2217/rme.15.85. Epub 2016 Feb 29. PMID 26925512
- [Background] Kurobe H, Tara S, Maxfield MW, Rocco KA, Bagi PS, Yi T, Udelsman BV, Dean EW, Khosravi R, Powell HM, Shinoka T, Breuer CK. Comparison of the biological equivalence of two methods for isolating bone marrow mononuclear cells for fabricating tissue-engineered vascular grafts. Tissue Eng Part C Methods. 2015 Jun;21(6):597-604. doi: 10.1089/ten.TEC.2014.0442. Epub 2014 Dec 29. PMID 25397868
- [Background] Kurobe H, Maxfield MW, Naito Y, Cleary M, Stacy MR, Solomon D, Rocco KA, Tara S, Lee AY, Sinusas AJ, Snyder EL, Shinoka T, Breuer CK. Comparison of a closed system to a standard open technique for preparing tissue-engineered vascular grafts. Tissue Eng Part C Methods. 2015 Jan;21(1):88-93. doi: 10.1089/ten.TEC.2014.0160. PMID 24866863
- [Background] Hibino N, McGillicuddy E, Matsumura G, Ichihara Y, Naito Y, Breuer C, Shinoka T. Late-term results of tissue-engineered vascular grafts in humans. J Thorac Cardiovasc Surg. 2010 Feb;139(2):431-6, 436.e1-2. doi: 10.1016/j.jtcvs.2009.09.057. PMID 20106404